CLINICAL TRIAL: NCT07088471
Title: Cardiac Left Atrial Evaluation and Response in HFrEF With Sacubitril/Valsartan: The CLEAR Study.
Brief Title: Cardiac Left Atrial Evaluation and Response in HFrEF With Sacubitril/Valsartan
Acronym: CLEAR
Status: Active, not recruiting | Type: Observational
Sponsor: Connolly Hospital Blanchardstown (Other)
Responsible Party: Principal Investigator, Michael J Daly, MA MD PhD, Dr, Connolly Hospital Blanchardstown
Other Study IDs: CHB 005/25
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure and Reduced Ejection Fraction
Keywords: left atrial strain; Sacubril/valsartan; HFrEF; Heart Failure
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure | interventions — Valsartan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Sacubtril/Valsartan — Angiotensin-receptor blocker and neprilysin inhibitor therapy

SUMMARY:
Heart failure is an increasingly common condition that can have a significant impact on quality of life and reduce life expectancy. In recent decades, a number of drugs have been developed specifically for this condition. One such drug, called Sacubitril/valsartan (SV) has been shown to reduce hospitalizations and prolong life expectancy of patients with heart failure. It works by reversing some of the structural and functional changes to the heart that occur in heart failure. However, not all patients respond to the drug. Further research is needed to better understand the reasons for this and predict who will benefit most from the drug.

Left atrial strain is a relatively new measurement that can be obtained using ultrasound imaging of the heart, and it provides objective information about how one of the heart's four chambers is functioning. The investigators aim to assess the effect of SV therapy on left atrial strain in patients with heart failure. The investigator's objective is to understand whether abnormal left atrial strain or changes in left atrial strain help predict response to SV therapy.

DETAILED DESCRIPTION:
Sacubitril/valsartan (SV) improves cardiovascular outcomes in patients with heart failure and reduced ejection fraction (HFrEF) [1]. However, not all patients respond to therapy. SV therapy has been shown to promote reverse cardiac remodelling, which may contribute to its efficacy in responders [2].

Left atrial (LA) remodeling has been shown to be related to a variety of cardiovascular diseases. Until recently, the LA was only considered to act as a conduit for the left ventricle, and we now know that the LA plays a dynamic role throughout the cardiac cycle. Currently, LA volume is recommended by the European Society of Cardiology for the evaluation of LA size and remodeling [2]. Over the last decade, advancements in echocardiographic software have led to the development of novel parameters to measure LA function and remodeling. LA function is now divided into three phases: reservoir, conduit, and contractile phase.

Recently, speckle tracking on 2-dimensional echocardiography has been used to evaluate LA Strain. LA strain has been evaluated in clinical studies and has been shown to be a useful tool in the diagnosis of LA remodeling when compared to conventional methods. A recently published study from Korea has defined the reference ranges for LA strain in a healthy population [3]. Along with the reference range, the same study also looked at different determinants of LA strain [3]. LA strain by speckle tracking echocardiography is an affordable, non-invasive, pragmatic, diagnostic tool that can be performed as part of the standard 2D echocardiogram.

There have been limited studies assessing the relationship between SV therapy and LA strain. The investigators aim to evaluate the hypothesis that baseline LA strain and any changes associated with SV therapy may be a prognosticator of response to therapy in HFrEF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults diagnosed with heart Failure with reduced ejection fraction (HFrEF), i.e. LVEF ≤40% by Simpson's method on transthoracic echocardiography
2. Stable guideline-directed medical therapy prior to sacubitril/valsartan (SV) initiation
3. New York Heart Association classes II-III symptom status
4. Guideline-directed up-titration of SV therapy to the maximum tolerated dose
5. Transthoracic echocardiogram and NT-proBNP prior to SV initiation and at 3 months post commencement of therapy

Exclusion Criteria:

1. Patients not in sinus rhythm at time of echocardiograms (precludes left atrial strain analysis)
2. Sub-optimal echocardiographic images to allow measurement of left atrial strain
3. Prior mitral valve intervention (left atrial strain assessment unreliable in this cohort)
4. Severe mitral regurgitation (left atrial strain assessment unreliable in this cohort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure with reduced ejection fraction (HFrEF) patients on stable guideline-directed medical therapy prior to commencing sacubitril/valsartan (SV) will be retrospectively identified
Sampling Method: Non-Probability Sample
Enrollment: 334 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between pre-therapy left atrial strain parameters on speckle-tracking echocardiography and therapy-associated changes in left ventricular ejection fraction and/or serum NT-pro BNP. | At least 3-6 months post initiation of SV therapy
  Correlation between baseline, pre-therapy left atrial strain parameters on speckle-tracking echocardiography (TTE) with therapy-associated changes in left ventricular ejection fraction (LVEF) on TTE and serum NT-pro BNP. LVEF will be assessed on TTE using the modified Simpson's biplane method. Left atrial strain will be assessed using speckle tracking analysis with EchoPAC Software v204 (GE Vingmed Ultrasound AS, Horten, Norway). Correlation will be assessed using Spearman's rank correlation coefficients.

SECONDARY OUTCOMES:
Correlation between pre-therapy left atrial strain parameters and baseline left ventricular ejection fraction and serum NT-pro BNP level. | At least 3-6 months post initiation of SV therapy
  Correlation between baseline left atrial strain values and baseline left ventricular ejection fraction and NT-pro BNP. LVEF will be assessed using the modified Simpson's biplane method. Left atrial strain will be assessed using speckle tracking analysis with EchoPAC Software v204 (GE Vingmed Ultrasound AS, Horten, Norway). Correlation will be assessed using Spearman's rank correlation coefficients.
Mean change in left atrial strain parameters pre- and post-SV therapy | At least 3-6 months post initiation of SV therapy
  Mean change in left atrial reservoir, conduit, and booster pump values pre- and post-SV therapy. Left atrial strain will be assessed using speckle tracking analysis with EchoPAC Software v204 (GE Vingmed Ultrasound AS, Horten, Norway).
Correlation between therapy-associated changes in left atrial strain parameters and therapy-associated changes in left ventricular ejection fraction and/or serum NT pro-BNP level. | At least 3-6 months post initiation of SV therapy
  Correlation between therapy-associated changes in left atrial strain and therapy-associated changes in left ventricular ejection fraction or NT pro-BNP. LVEF will be assessed using the modified Simpson's biplane method. Left atrial strain will be assessed using speckle tracking analysis with EchoPAC Software v204 (GE Vingmed Ultrasound AS, Horten, Norway). Correlation will be assessed using Spearman's rank correlation coefficients.

CONTACTS AND LOCATIONS:
Locations (1):
- Connoly Hospital Blanchardstown, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Data can be made available upon reasonable request